CLINICAL TRIAL: NCT04760379
Title: Effect of Focal Muscle Vibration on Flexibility and Perceived Stiffness in Patients With Mechanical Low Back Pain
Brief Title: Focal Muscle Vibration on Flexibility and Perceived Stiffness in Patients With Mechanical Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00906 Maham Malik
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Active Comparator): Bridging, Stretching exercises (quadratus lumborum, erector spinae) McKenzie exercises and TENS (10 mins).
  Interventions: Other: Conventional therapy
- Vibration Therapy (Experimental): Focal muscle vibrator (FMV) (120 Hz) for 10 minutes on paraspinal muscles. Bridging, Stretching exercises (quadratus lumborum, erector spinae) McKenzie exercises and TENS (10 mins).
  Interventions: Other: vibration therapy

INTERVENTIONS:
Other: Conventional therapy — Bridging, Stretching exercises (quadratus lumborum, erector spinae) McKenzie exercises and TENS (10 mins).
  Arms: Conventional Therapy
Other: vibration therapy — Focal muscle vibrator (120 Hz) for 10 minutes on paraspinal muscles. Bridging, Stretching exercises (quadratus lumborum, erector spinae) McKenzie exercises and TENS (10 mins).
  Arms: Vibration Therapy

SUMMARY:
Low back pain that does not have any known specific pathology i.e.: tumor, any infection, fracture, osteoporosis, structural deformity, radicular syndrome, inflammatory disorder or cauda equine syndrome) is referred as non-specific low back pain.Over worldwide low back pain is a major public health challenge. Low back pain prevalence is shown to be 84% while 23% of chronic low back pain. Disability due to low back pain is about 11 to 12%. Low back pain is a leading cause of increasing economic burden in respect to huge medical expenses. Statistical analysis of indirect and direct expenses for the low back pain treatment in U.S shows over $100 billion per year.Many risk factors for low back pain has been identified including degeneration of lumbar discs, over weight/obesity, sedentary life style and mechanical factors i.e. occupational sitting, manual handling and assisting patients, awkward postures, lifting and carrying weights. Exercise therapy is suggested as an effective treatment in improving function of the back muscles and relieving pain in patients with Low back pain. Many studies suggested that muscle vibration is effective as the vibration signals are delivered via an external stimulator that is exposed to the part of the body resulting in pain relief and reducing muscle spasm. Vibratory stimuli have practical uses in rehabilitation and in exercise performance. Increasing reflexive activity through the stimulation of muscle spindles results in tonic vibratory reflex. The mechanical and electrical responses of the muscle could vary with the frequency of the vibration to the muscle. LMV effects are localized to the point where the stimulation is given and this is the result of neurogenic potentiation through the tonic vibratory reflex from the stimulation of muscle spindles. In our study we will work with 120hz frequency to improve the flexibility and perceived stiffness.

DETAILED DESCRIPTION:
Evidence suggests that a period of localized muscle stimulation have positive effects on muscle function and in relieving pain and muscular stiffness.

In 2014 local muscle vibration frequency's acute effects on peak torque, EMG activity and rate of torque development was studied. The purpose of this study was to examine the effects of vibration on quadriceps muscle. Findings of this study suggest that local muscle vibration can encourage improvement in quadriceps activation and it can be useful in the treatment of quadriceps dysfunction that can occur in several knee pathologies.

A study was conducted in 2009 to examine the effects of vibration on arm muscles during isometric activity of muscles. Analysis according to the recordings revealed a significant increase in the waves on electromyography when vibration was applied. This study results revealed that vibration given to the specific muscles produces an increase of the activation and the coactivation.

A study in 1999 was held to investigate the effects of muscle vibration on the muscle spindles of Para spinal muscles in active lumbosacral position sense in sitting .This study suggest that muscle vibration technique was used to alter the potential afferent input from these Para spinal muscle receptors. Result shows that the muscle vibration on multifidus encouraged the illusion of significant muscle lengthening in the patients.

Another study in 2003 was held to inspect the facilitation of triceps brachii muscle contraction by applying the vibration on tendon after chronic cervical spinal cord injury. The efficacy of the vibration was checked by the analysis of a tonic vibration reflex was induced in each of the triceps brachii muscles at rest. If a reflex response was induced by the vibration before or during the voluntary contraction of the triceps brachii, vibration may facilitate the initiation, maintenance, and/or strength of the voluntary contraction.

ELIGIBILITY:
Inclusion Criteria:

• Having mechanical low back pain from past 3 months

Exclusion Criteria:

* Patients with neurological symptoms
* Back operations 6 months before
* Leg length discrepancies
* Those diagnosed with bony deformity of spine like scoliosis and spondylolisthesis.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sit and Reach Test | Change from baseline to 4 weeks
  The sit and reach test is the most common of all flexibility tests. It measures the flexibility of the clients' lower back and hamstrings. All you need is a box about 30cm high and a meter ruler.
  * Your client should sit on the floor with their back and head against a wall. Their legs should be out straight ahead and their knees flat against the floor.
  * Place the box against your client's feet (no shoes). Whilst keeping their head and back against the wall, instruct your client to stretch out their arms as far as they can towards the box without their head or back loosing contact with the wall.
  * Place the ruler on the box and move the zero end towards your clients fingertips. When the ruler touches their fingertips you have the zero point and the test can begin.
  * Instruct your client to lean forward slowly as far as possible keeping their fingertips level with each other and their legs flat on the floor. Their head and shoulders can come away from the wall now.
  * Slowly
Likert stiffness scale: | Change from baseline to 4 weeks
  this is 7 points scale, o indicate a complete absence of soreness and 6 indicates a severe muscle soreness,stiffness and weakness that limits my ability to move

SECONDARY OUTCOMES:
Numeric Pain Rating Scale: | Change from baseline to 4 weeks
  General Information:
  * The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours.
  * The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours.
    • Patient Instructions (adopted from (McCaffery, Beebe et al. 1989):
  * "Please indicate the intensity of current, best, and worst pain levels over the past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable)"

CONTACTS AND LOCATIONS:
Overall Officials: Anam Qureshi, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang XQ, Pi YL, Chen PJ, Chen BL, Liang LC, Li X, Wang X, Zhang J. Whole body vibration exercise for chronic low back pain: study protocol for a single-blind randomized controlled trial. Trials. 2014 Apr 2;15:104. doi: 10.1186/1745-6215-15-104. PMID 24693945
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Pamukoff DN, Ryan ED, Blackburn JT. The acute effects of local muscle vibration frequency on peak torque, rate of torque development, and EMG activity. J Electromyogr Kinesiol. 2014 Dec;24(6):888-94. doi: 10.1016/j.jelekin.2014.07.014. Epub 2014 Aug 7. PMID 25169762
- [Background] Mischi M, Cardinale M. The effects of a 28-Hz vibration on arm muscle activity during isometric exercise. Med Sci Sports Exerc. 2009 Mar;41(3):645-53. doi: 10.1249/MSS.0b013e31818a8a69. PMID 19204585
- [Background] Brumagne S, Lysens R, Swinnen S, Verschueren S. Effect of paraspinal muscle vibration on position sense of the lumbosacral spine. Spine (Phila Pa 1976). 1999 Jul 1;24(13):1328-31. doi: 10.1097/00007632-199907010-00010. PMID 10404575